CLINICAL TRIAL: NCT05559606
Title: An Observational Study to Evaluate the Safety and Efficacy of Fixed Dose Combination Therapy With Atorvastatin and Ezetimibe in Real World Patients With Primary Hypercholesterolemia
Brief Title: An OS to Evaluate the Safety & Efficacy of Fixed Dose Combination Therapy With Atorvastatin and Ezetimibe
Acronym: LITE
Status: Completed | Type: Observational
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: BR-EAC-OS-401
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Primary Hypercholesterolemia
Keywords: Hypercholesterolemia; Atorvastatin; Ezetimibe
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study observes real world patients with primary hypercholesterolemia who receive a fixed dose combination therapy with atorvastatin and ezetimibe for 24 weeks; collects and analyzes data related to efficacy and safety of the therapy; and evaluates efficacy and safety of the fixed dose combination therapy with atorvastatin and ezetimibe.

DETAILED DESCRIPTION:
The prevalence of hypercholesterolemia, an atherosclerotic dyslipidemia which is the major cause of coronary artery diseases has risen. According to numerous studies, LDL-C is the key cause of atherosclerosis and it has been reported that treating patients to lower the LDL-C level will reduce the incidence of cardiovascular diseases. Currently, patients are classified into risk groups to receive a recommended therapy based on the defined criteria in Korea and Statin is the primary therapeutic agent recommended. However, there have been concerns that an increased dose of statins may result in hepatoxicity and reports that a combination therapy with ezetimibe without an additional dose of statins has clinical benefits. Ezetimibe is a drug that inhibits cholesterol absorption in the small intestine and reduces the LDL-C level. The therapeutic guideline, first of all, recommends combination therapy with ezetimibe among other drugs whose clinical benefits have been confirmed in cases where the target LDL-C level is not met with statins.

The study observes real world patients with primary hypercholesterolemia who receive a fixed dose combination therapy with atorvastatin and ezetimibe for 24 weeks; collects and analyzes data related to efficacy and safety of the therapy; and evaluates efficacy and safety of the fixed dose combination therapy with atorvastatin and ezetimibe.

During this study period, the scope of data to be collected is as follows:

* Demographic data
* Indication diagnosis and characteristics
* Cardiovascular risk
* Medical history
* Statin medication
* Preceding/Concomitant drug
* Administration of fixed dose combination therapy with atorvastatin and ezetimibe
* Collecting efficacy endpoints: Lipid profile(LDL-C, TC, TG, HDL-C, non-HDL-C)
* Collecting safety endpoints: ADR, SAE, SADR, HbA1C, FPG, AST, ALT, CPK

ELIGIBILITY:
Inclusion Criteria:

1. Those who are briefed about the clinical trial objectives and methods, and express their consent to participate in the trial by signing a written consent on the use of their personal information.
2. Any male/female subjects 19 years old or older.
3. Those who will be given for the first time a fixed dose combination therapy with atorvastatin and ezetimibe to treat primary hypercholesterolemia.
4. Those with levels of total cholesterol, LDL-C, HDL-C, non-HDL-C and TG confirmed within 2 weeks prior to the registration.
5. Those who failed to reach to the target LDL-C level per risk group based on the risk group classification specified in the therapeutic guideline for dyslipidemia (2018).

   [Risk Group, Target LDL-C (mg/dL) Level]
   * Very High Risk <70

     * Coronary artery disease
     * Atherosclerotic ischemic stroke and transient cerebral ischemic attack
     * Peripheral arterial disease
   * High Risk <100

     * Carotid disease (When significant carotid artery stenosis is diagnosed)
     * Abdominal aneurysm
     * Diabetes (For patients with major risk factors such as damage to target organs or cardiovascular diseases, the target level may be lowered based on the patient conditions)
   * Moderate Risk <130

     * 2 or more major risk factors(May include age (45 years old for male subjects and 55 years old for female subjects), family history of initial coronary artery disease stage, hypertension, smoking, low HDL-C)
   * Low Risk <160

     * 1 or less major risk factors(May include age (45 years old for male subjects and 55 years old for female subjects), family history of initial coronary artery disease stage, hypertension, smoking, low HDL-C)
6. Those who fully understand the clinical trial, are cooperative throughout the trial and capable of participating in the trial until it ends.

Exclusion Criteria:

1. Those who are hypersensitive to major ingredients or other ingredients of the investigational drug.
2. Hypertriglyceridemia patients whose triglyceride level is 400mg/dL or higher under fasting conditions.
3. Patients with serious hepatopathy (whose ALT or AST level is more than twice the upper limit of normal (ULN)).
4. Patients with serious nephropathy.
5. Those who have medical history of myopathy and rhabdomyolysis.
6. Female patients who are pregnant, suspected to be pregnant or breastfeeding.
7. Those who are administrating glecaprevir and pibrentasvir.
8. The drug contains lactose, thus those who have genetic problems, including galactose intolerance, Lapp lactase deficiency and glucose-galactose malabsorption.
9. Those who are currently participating in other clinical trials (any trials with drugs or medical devices) or who have been administered with investigational drugs of other clinical trials within 4 weeks from the baseline. However, those participating in non-interventional trials or being observed after the drug administration is complete may take part in the trial.
10. Those who are currently hospitalized or are expected to be hospitalized.
11. Those who are suffering from severe or unstable medical and mental illnesses that may impact the trial as assessed by the investigators.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary hypercholesterolemia that require a fixed dose combination therapy with Atorvastatin and Ezetimibe
Sampling Method: Non-Probability Sample
Enrollment: 1839 (Actual)
Dates: Start 2022-09-07 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Rate of reaching the target LDL-C level | Week 24
  Rate of reaching the target LDL-C level at Week 24

SECONDARY OUTCOMES:
Rate of reaching the target LDL-C level | Week 12
  Rate of reaching the target LDL-C level at Week 12
Rate of change compared to the baseline when it comes to the level of TC, TG, LDL-C, HDL-C and non-HDL-C | Week 12 and Week 24
  Rate of change at Week 12 and Week 24 compared to the baseline when it comes to the level of TC, TG, LDL-C, HDL-C and non-HDL-C

CONTACTS AND LOCATIONS:
Overall Officials: MyungSook Hong, Study Director — Boryung Co.,Ltd.
Locations (1):
- Severance Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No